CLINICAL TRIAL: NCT06901076
Title: Effect of a Food Supplement Based on Nigella Sativa Seeds Oil and Vitamin E on Glyco-lipid Parameters in Dysglycemic and Dyslipidemic Perimenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NST 01
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Perimenopausal Disorder; Impaired Glucose Tolerance; Impaired Fasting Glycemia
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: Two-arm randomized, placebo-controlled, double-blind, parallel-groups trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nisatol (Experimental): Nisatol® (developed by PharmExtracta) containing Nigella sativa seeds oil and Vitamin E, 1 capsule soft gel after breakfast and 1 capsule soft gel after dinner for 6 months
  Interventions: Dietary Supplement: Nisatol
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nisatol — Nisatol® (developed by PharmExtracta) containing Nigella sativa seeds oil and Vitamin E, 1 capsule soft gel after breakfast and 1 capsule soft gel after dinner for 6 months
  Arms: Nisatol
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A total of 120 subjects in one center will be enrolled and will be divided into two treatment groups of 60 subjects each with 1:1 allocation ratio. Permuted block randomization will be used. Active treatment inlcude Nisatol® (developed by PharmExtracta) containing Nigella sativa seeds oil and Vitamin E, 1 capsule soft gel after breakfast and 1 capsule soft gel after dinner for 6 months; Control Intervention is Placebo.

DETAILED DESCRIPTION:
In the screening visit subject's demographic data, medical history, comorbidities and concomitant medication will be collected. Patients who are dysglycemic following OGTT and who are also dyslipidemic will be evaluate. Blood sample analysis will be prescribed to be performed before the next visit for the evaluation of FPG, FPI, TC, HDL-C, Tg, ALT, AST, uric acid, creatinine, lipoprotein(a) [Lp(a)], high sensitive C-reactive protein (hs-CRP), 25-hydroxyvitamin D3 (25-OH D3), follicle stimulating hormone (FSH), estradiol, androstenedione, dehydroepiandrosterone sulphate (DHEAS), cortisol, thyroid stimulating hormone (TSH). Blood sample analysis will be performed in amenorrhea or within the first 3 days of the menstrual cycle. Adiponectin (ADN), resistin, oxidized LDL (oxLDL) and malondialdehyde (MDA) will be assessed by using enzyme-linked immunosorbent assay (ELISA) kits commercially available. At the baseline visit, a 12-lead ECG will be recorded to exclude ischemic disease and a computerized medical record will be compiled where the following data will be recorded: vital signs [waist circumference, abdomen circumference, hip circumference, weight, height, body mass index (BMI), systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR)] the laboratory tests (FPG, FPI, TC, HDL-C, Tg, ALT, AST, uric acid, creatinine, Lp(a), hs-CRP, 25-OH D3, FSH, estradiol, androstenedione, DHEAS, cortisol, TSH) and the parameters detected with ELISA kits (ADN, resistin, oxLDL and MDA). There will be calculated LDL-C and homeostasis model assessment of insulin resistance (HOMA-IR). Perimenopausal symptoms were assessed using WHQ and estrogen-androgenic climacteric syndrome questionnaires. In addition anxiety and depression were evaluated in perimenopausal women with the HADS. The female sexual function index and the FSDS were used for the measurement of sexual function and distress. The perimenopausal women will be randomized in one of the 2 groups to receive the food supplement or placebo and a sufficient amount of study product for 6 months will be delivered. All subjects will receive dietary recommendations. After 3 months of treatment vital signs will be recorded. The Investigator will verify the product tolerability. Any adverse events eventually occurred will be collected. Perimenopausal symptoms were assessed using WHQ and estrogen-androgenic climacteric syndrome questionnaires. In additionanxiety and depression were evaluated in perimenopausal women with the HADS. The female sexual function index and the FSDS were used for the measurement of sexual function and distress. Blood sample analysis will be prescribed to be performed before the next visit for the evaluation of FPG, FPI, TC, HDL-C, Tg, ALT, AST, uric acid, creatinine, Lp(a), hs-CRP, 25-OH D3, FSH, estradiol, androstenedione, DHEAS, cortisol, TSH. After 6 months of treatment, following blood samples collection, the perimenopausal women will be undergone to an OGTT to reevaluate the dysglycemia status at the end of the study; laboratory tests and the parameters detected with ELISA kits will be recorded. There will be calculated LDL-C and HOMA-IR. The Investigator will verify the product tolerability. Any adverse events eventually occurred will be collected. Perimenopausal symptoms were assessed using WHQ and estrogenandrogenic climacteric syndrome questionnaires. In addition anxiety and depression were evaluated in perimenopausal women with the HADS. The female sexual function index and the FSDS were used for the measurement of sexual function and distress.

ELIGIBILITY:
Inclusion Criteria:

* perimenopausal women (irregular cycles up to intervals of more than 60 days)
* FPG values between 100 and 125 mg/dl and confirmation with oral glucose tolerance test (OGTT)
* TC values ≥ 200 mg/dl

Exclusion Criteria:

* neoplastic diseases
* liver diseases
* renal insufficiency
* diabetes mellitus

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Effect on cholesterol and glycemia | 6 months
  The primary outcome is the comparison of two arms (Nisatol® supplement vs Placebo) for the effects on fasting plasma glucose and total cholesterol

SECONDARY OUTCOMES:
LDL and HDL-cholesterol | 6 months
  Effetcs of the two treatments on LDL-Cholesterol and HDL-Cholesterol
Glycemic status | 6 months
  Proportion of perimenopausal women passing from impaired fasting glucose condition to euglycemia; from impaired glucose tolerance condition to euglycemia; from impaired fasting glucose condition to diabetes; from impaired glucose tolerance condition to diabetes

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Medicina Generale 1, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be presented and discussed in an original article